CLINICAL TRIAL: NCT01495156
Title: A Randomized, Double-blind, Placebo Controlled Study of the Efficacy of Adjunctive Lithium for the Treatment of Psychotic Mania Followed by an Open Label Long-term Safety Period.
Brief Title: Study of the Efficacy of Adjunctive Lithium Treatment for the Treatment of Psychotic Mania
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-185
Record Dates: First submitted 2011-11-22; First posted 2011-12-19 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Bipolar I Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lithium/Adjunctive SGA (Experimental)
  Interventions: Drug: Lithium treatment in combination with a SGA (Second Generation Antipsychotic)
- Placebo/Adjunctive SGA (Placebo Comparator)
  Interventions: Drug: Placebo/Adjunctive SGA treatment

INTERVENTIONS:
Drug: Lithium treatment in combination with a SGA (Second Generation Antipsychotic) — All patients will be treated with aripiprazole with a target dose of 10 mg/day and a max daily dose of 30 mg. If aripiprazole is ineffective or not tolerated, it will be tapered and risperidone treatment will be started. If patient had an adequate aripiprazole trial in the past as described above, risperidone will be the initial treatment. Risperidone dosing will begin with 0.5 mg/day on day 1 with a target dose of 2.5 mg/day and a max daily dose of 6mg.
  Subjects in the lithium /adjunctive SGA group will be started at 900 mg/day lithium in thrice daily dosing. The lithium dose will be increased to 1200mg/day on day 4 if lithium has been well-tolerated and symptoms of mania remain, as determined by a phone assessment done by a blinded study physician. The target serum level of lithium will be 1.2 mEq/L (range 0.8 to 1.4 mEq/L).
  Arms: Lithium/Adjunctive SGA
Drug: Placebo/Adjunctive SGA treatment — All patients will be treated with aripiprazole with a target dose of 10 mg/day and a max daily dose of 30 mg. If aripiprazole is ineffective or not tolerated, it will be tapered and risperidone treatment will be started. If patient had an adequate aripiprazole trial in the past as described above, risperidone will be the initial treatment. Risperidone dosing will begin with 0.5 mg/day on day 1 with a target dose of 2.5 mg/day and a max daily dose of 6mg.
  Subjects in the placebo /adjunctive SGA group will receive placebo for the entire trial in addition to the adjunctive SGA.
  Arms: Placebo/Adjunctive SGA

SUMMARY:
The proposed pilot study is a placebo-controlled, parallel group, randomized clinical trial comparing two treatment strategies in adolescents with mania and prominent psychotic features. One group will receive a second generation antipsychotic (SGA) and placebo and the other will receive a SGA and lithium.

The primary double-blind phase of the study will last 8 weeks, followed by a 24-week extension-phase.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 12-18 years old, inpatients or outpatients
* meet DSM-IV criteria for Bipolar I disorder - manic or mixed episode
* psychotic symptoms present

Exclusion criteria:

* current serious homicidal/suicidal ideation
* prior non-response or intolerance to an adequate trial of lithium
* prior non-response or intolerance to adequate trials of both aripiprazole and risperidone
* any unstable medical condition or medical contraindication to treatment with lithium, aripiprazole or risperidone
* inability or unwillingness to discontinue concomitant medication that interferes with the pharmacokinetics of either lithium, aripiprazole, or risperidone
* seizure disorder
* pregnant or, if sexually active, not using birth control, such as oral contraceptives, two barrier methods, long-acting depot preparations or an intra-uterine device
* Full Scale IQ less than 70
* meets criteria for a DSM-IV diagnosis of substance-induced mood disorder or mood disorder due to a general medical condition.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2014-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Acute phase :Time to partial or full response | 8 weeks
  Acute phase: Partial response is defined as at least a 25% -49% reduction in YMRS score and a CGI improvement item score of 2. Full response is defined as a reduction in YMRS score of 50% or more and a CGI improvement item score of 1 "very much improved."
Continuation Phase: time to recurrence of a subsyndromal mood episode | 24 weeks
  We will measure the amount of time for patients to have a recurrance of a subsyndomal mood episode during the Continuation Phase

SECONDARY OUTCOMES:
Acute phase: number of suicidal events | 8 weeks
Acute phase: positive urine toxicology screens (yes/no variable) | 8 weeks
Acute phase: adherence to medication regimen. | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Zucker Hillside Hospital, North Shore-LIJ Health System, Glen Oaks, New York, United States